CLINICAL TRIAL: NCT04036396
Title: Mobile Enhanced Prevention Support for People Leaving Jail
Acronym: MEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles Centers For Alcohol and Drug Abuse (Unknown); Charles Drew University of Medicine and Science (Other); California HIV/AIDS Research Program (Other); Friends Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Nina T. Harawa, MPH, PhD, Professor-in-Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-000165; OS17-LA-003 (Other Grant/Funding Number: California HIV/AIDS Research Program)
Record Dates: First submitted 2019-03-29; First posted 2019-07-29 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections; Sexually Transmitted Diseases, Bacterial; Hepatitis C; Substance Use Disorders
Keywords: HIV prevention and testing; sexually transmitted disease (STD) prevention and testing; HIV pre-exposure prophylaxis (PrEP); Incarceration
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases, Bacterial; Hepatitis C; Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: The Mobile Enhanced Prevention Support (MEPS) intervention is designed to support, motivate, and facilitate engagement in preventive health care activities in the period of community reentry following jail. Three components: support from a selected Peer Mentor (PM), incentives, and a developed mobile application. Client-driven approach, in which participants are encouraged to address priorities and immediate needs for that they identify a client-centered needs assessment, prioritization, and wellness planning process, especially social determinants of health that may discourage or undermine preventive health measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): A client-centered assessment of priorities and needs and customized prevention and testing referrals.
  Interventions: Behavioral: Usual Care plus Customized Referrals
- Mobile Enhanced Prevention Support (Experimental): Standard of Care in addition to a client-centered assessment of priorities and needs and customized prevention and testing referrals, and the Mobile Enhanced Prevention Support Program
  Interventions: Behavioral: Mobile Enhanced Prevention Support; Behavioral: Usual Care plus Customized Referrals

INTERVENTIONS:
Behavioral: Mobile Enhanced Prevention Support — Access to the newly developed GeoPassport App, incentives for accessing identified services, and a trained Peer Mentor.
  Other Names: MEPS
  Arms: Mobile Enhanced Prevention Support
Behavioral: Usual Care plus Customized Referrals — Participants in the control arm will continue to receive services they would normally receive consistent with the setting in which they were recruited. This includes substance use treatment in jail, substance use treatment at a residential recovery facility, and/or supportive housing services. The study will provide referrals customized to their needs and preferences.

SUMMARY:
This study will provide HIV prevention and related support services to men who have sex with men and transgender women who have substance use disorders and are either leaving jail or recently released from jail. The researchers will compare the utilization of HIV prevention and other support services between individuals who receive routine case management provided following enrollment to those who have access to GeoPassport, a global position service (GPS)-based mobile app, incentives, and peer mentor support.

DETAILED DESCRIPTION:
The investigators will enroll 200 people in jail or within 12 months post-release from incarceration. During the trial, half of participants will be randomized into a control group that will receive usual care consistent with the setting in which they live, along with referrals customized to their needs and preferences to share with a case manager. They will be compared to the other half of participants randomized to the intervention group that, in addition to receiving customized referral sources, will also receive the GeoPassport App, incentives, and the support of a trained Peer Mentor for six months. The GeoPassport App will provide participants with tools for tracking goals and progress toward meeting them, assistance in locating services, appointment and medication reminders, opportunities to provide feedback on service providers, and built-in tracking and distribution of rewards (incentives) for service utilization. GeoPassport will assist Peer Mentors in monitoring participants' service utilization. The Peer Mentors will provide encouragement, role modeling, accompaniment to appointments, and assistance with goal setting, problem-solving, and reducing logistical and psychosocial barriers to service engagement. The intervention can be delivered in person or remotely in order to comply with necessary social distancing during the COVID-19 pandemic. Participants in both groups will be followed to assess whether those offered the intervention are more likely to meet the specific prevention targets described in the Specific Aims. The intervention lasts 6 months from the start of participation. Participants are interviewed at 3, 6, and 9 months from the same point as the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. housed in K6G unit or within 12 months post-release from incarceration
2. ages 18-49 years
3. screens positive for Substance Use Disorder (SUD), or has sought or received SUD treatment at any time starting 12 months before the most recent incarceration until the present day.
4. reports sexual intercourse with a male or a male-to-female transgender woman in the six months prior to jail entry
5. if recruited in jail, is likely to be remain either in custody for at least four more days, but less than three more months based on scheduled court dates, current sentence, treatment plan, etc.
6. has not received an HIV diagnosis (based on self-report)
7. plans to reside in Los Angeles County for the 12 months following enrollment

Exclusion Criteria:

1. does not have a smartphone and is not willing to obtain one post-release,
2. is not able to speak and understand English, and
3. does not have sufficient reading skills to operate a mobile app

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identifies as a man or a male-to-female trans woman.
Enrollment: 233 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina T Harawa, PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - God's Property, Los Angeles, California
  - Los Angeles County Men's Central Jail, Los Angeles, California
  - Los Angeles Center for Alcohol and Drug Abuse, Santa Fe Springs, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schrode KM, Edwards GG, Moghanian B, Weiss RE, Reback CJ, McWells C, Hilliard CL, Harawa NT. Randomized Controlled Trial Testing an HIV/STI Prevention Intervention Among People Leaving Incarceration Who Were Assigned Male at Birth, Have Sex with Men and A Substance Use Disorder. AIDS Behav. 2025 Dec;29(12):3806-3821. doi: 10.1007/s10461-025-04818-4. Epub 2025 Jul 10. PMID 40634829
- [Derived] Edwards GG, Reback CJ, Cunningham WE, Hilliard CL, McWells C, Mukherjee S, Weiss RE, Harawa NT. Mobile-Enhanced Prevention Support Study for Men Who Have Sex With Men and Transgender Women Leaving Jail: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 22;9(9):e18106. doi: 10.2196/18106. PMID 32959786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a variety of methods, including direct recruitment at supportive housing facilities in LA County and in MCJ, referrals from community partners, participant referrals, and flyers posted by community organizations.
Period: Overall Study
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Started | 117 | 116
Completed | 86 | 87
Not Completed | 31 | 29
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 12 | 14
Not completed — Determined ineligible after enrollment | 14 | 10

BASELINE CHARACTERISTICS:
Population: Participants who were enrolled and began the study but were later determined to be ineligible are excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (7.6) | 32.5 (6.6) | 33.5 (7.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender identity: Cisgender male | 90 | 88 | 178
  Gender identity: Trans female | 8 | 11 | 19
  Gender identity: Gender non-binary or non-conforming | 4 | 5 | 9
  Gender identity: Other | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: American Indian or Alaska Native | 1 | 1 | 2
  Race/ethnicity: Asian | 2 | 2 | 4
  Race/ethnicity: Black or African American | 26 | 27 | 53
  Race/ethnicity: Hispanic or Latino | 47 | 40 | 87
  Race/ethnicity: Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  Race/ethnicity: White | 18 | 26 | 44
  Race/ethnicity: Other (usually multiple) | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 103 | 105 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Establishing a Primary Care Provider Who Can Prescribe PrEP (Pre-exposure Prophylaxis)
Description: Defined as the participant identifying and completing an appointment with a primary care provider who is willing and able to prescribe HIV pre-exposure prophylaxis.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 93 | 99
Participants | 82 | 90
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.780, Poisson regression; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.66 to 1.74]

2. Primary Outcome: Number of Participants Who Initiate PrEP Regimen
Description: Defined as the participant obtaining a prescription for PrEP, providing documentation, reporting taking the medication
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 86 | 87
Participants | 12 | 28
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.0006, Longitudinal trajectory model; Odds Ratio (OR) = 3.8, 95% CI 2-sided [1.8 to 8.0]

3. Primary Outcome: Number of Participants Who Demonstrate Minimal Adherence to PrEP
Description: Defined as the participant self-reporting taking prescribed PrEP at least 4 days per week at first instance of reporting taking PrEP
Time Frame: 3, 6, or 9 months
Population: Sample is based on the number of people who reported taking PrEP (14 for Standard of care; 28 for MEPS) but excludes those who declined to respond to the adherence question.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 11 | 26
Participants | 10 | 26
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.1191, Chi-squared

4. Primary Outcome: Number of Participants Who Remain on PrEP for at Least 3 Months.
Description: The outcomes is defined by self-reported PrEP use for 3 or more months
Time Frame: 9 months
Population: Sample is based on the number of people who reported taking PrEP (14 for Standard of care; 28 for MEPS) but excludes those who declined to respond to the this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 11 | 27
Participants | 7 | 17
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.9689, Chi-squared

5. Primary Outcome: Number of Participants Who Report an HIV Test Within 3 Months of a Follow-up
Description: Defined as the participant self-reporting having obtained HIV testing within 3 months of the follow-up
Time Frame: 3, 6, and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 84 | 86
Participants
  3 months | 44 | 55
  6 months | 32 | 50
  9 months | 31 | 33
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.1683, Mixed Models Analysis — 3 month follow-up
Statistical Analysis 2: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.0158, Mixed Models Analysis — 6 month follow-up
Statistical Analysis 3: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.6910, Mixed Models Analysis — 9 month follow-up

6. Primary Outcome: Number of Participants Who Undergo a Test for Gonorrhea, Syphilis, and Chlamydia Within 6 Months of a Follow-up
Description: Defined by the participant self-reporting having obtained testing for these sexually transmitted diseases (STDs) within the 6 months prior to a follow-up over the 9 month follow-up period
Time Frame: 6 and 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 78 | 76
Participants
  3 months | 33 | 41
  6 months | 32 | 40
  9 months | 28 | 29
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.5367, Mixed Models Analysis — 3 month follow-up
Statistical Analysis 2: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.3976, Mixed Models Analysis — 6 month follow-up
Statistical Analysis 3: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.9283, Mixed Models Analysis; 9 month follow-up

7. Primary Outcome: Number of Participants Who Undergo a Test for Hepatitis C
Description: Defined by the participant self-reporting having obtained at least one test for Hepatitis C
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 93 | 99
Participants | 80 | 85
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.620, Poisson regression; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.73 to 1.72]

8. Primary Outcome: Number of Participants Obtaining Treatment for Substance Use Disorders (SUDs) in the Community
Description: Defined by the participant self-report of completing SUD appointments within the 3 months following enrollment
Time Frame: 3 months
Population: Sample based on the first 3-month followup and excluding participants who skipped the question
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 84 | 86
Participants | 25 | 23
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = .6621, Chi-squared

9. Primary Outcome: Number of Participants Who Remain Engaged in Treatment for Substance Use Disorders (SUDs) in the Community,
Description: Defined by the participant self-reporting remaining engaged in treatment (i.e., continuing to attend meetings, counseling or other treatment activities) in the 3 months prior to the final follow-up interview.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 86 | 87
Participants | 11 | 4
Statistical Analysis 1: Comparison: Standard of Care vs Mobile Enhanced Prevention Support; Test type: Superiority; p = 0.0635, Fisher Exact

10. Secondary Outcome: Number of Participants in Each Arm Receiving Care and Treatment for Newly Diagnosed HIV or HCV Infections.
Description: Self-report of whether or not participants received follow-up care and treatment for HIV or hepatitis C infections diagnosed during study follow-up (n=200)
Time Frame: 3, 6, or 9 months
Population: Outcome is among those who acquired HIV or HCV during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 4 | 4
Participants | 2 | 3

11. Secondary Outcome: Number of Participants Who Recidivate
Description: Measure the comparative effectiveness of each intervention arm on reducing recidivism (n=200), quantified as the number of respondents who are reincarcerated.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 93 | 99
Participants | 29 | 35

12. Secondary Outcome: Number of Reincarcerations Among Those Who Recidivate
Description: Measure the comparative effectiveness of the intervention reducing recidivism (n=200), quantified as total number of reincarcerations over the study period among those who recidivate.
Time Frame: 9 months
Population: Outcome is among those who were reincarcerated at some point during the study.
Measure: Median (Inter-Quartile Range); unit: reincarcerations
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
Number analyzed (Participants) | 29 | 35
reincarcerations | 1 [1 to 2] | 2 [1 to 2]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Standard of Care | Mobile Enhanced Prevention Support
All-Cause Mortality (participants affected / at risk) | 2/103 | 2/106
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/106
Other Adverse Events (participants affected / at risk) | 0/103 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04036396/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04036396/SAP_001.pdf